CLINICAL TRIAL: NCT03290313
Title: a Randomized, Double Blind, Placebo-controlled, Multicenter Clinical Trial of Efficacy and Safety of Shu Gan yi Yang Capsule in the Treatment of Depression Associated With Erectile Dysfunction (Stagnation of Liver qi and Kidney Deficiency)
Brief Title: Clinical Trial Scheme of Shu Gan yi Yang Capsule
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Collaborators: Guizhou Yi Bai Pharmaceutical Co., Ltd. (Unknown); Peking University Sixth Hospital (Other); Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Jie Zhang,BD, Chief physician, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHZD-SGYY
Record Dates: First submitted 2017-08-22; First posted 2017-09-21 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Depression With Erectile Dysfunction
Keywords: Depression; erectile dysfunction; shu gan yi yang
MeSH Terms: conditions — Depression; Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shu gan yi yang capsule (Experimental): 4 capsules / time, 3 times / day, taking 8 weeks
  Interventions: Drug: shu gan yi yang capsule; Other: Supportive psychotherapy
- shu gan yi yang capsule capsule simulation agent (Placebo Comparator): 4 capsules / time, 3 times / day, taking 8 weeks
  Interventions: Drug: shu gan yi yang capsule simulation agent; Other: Supportive psychotherapy

INTERVENTIONS:
Drug: shu gan yi yang capsule — Patients who did not use any antidepressants were given normal clinical medication； Patients who have been treated with antidepressants have been treated for more than 1 month and have reached a therapeutic dose without having to adjust the drug and dose within 2 months.In the original treatment on the basis of the same type of load to the clinical trial medication
  Arms: shu gan yi yang capsule
Drug: shu gan yi yang capsule simulation agent — Patients who did not use any antidepressants were given normal clinical medication； Patients who have been treated with antidepressants have been treated for more than 1 month and have reached a therapeutic dose without having to adjust the drug and dose within 2 months.In the original treatment on the basis of the same type of load to the clinical trial medication
  Arms: shu gan yi yang capsule capsule simulation agent
Other: Supportive psychotherapy — Each patient was given cognitive behavioral adjustment and supportive psychotherapy during the clinical trial

SUMMARY:
Shu gan yi yang capsule is made of traditional Chinese medicine Guizhou Yi Bai pharmaceutical Limited by Share Ltd, for liver and kidney deficiency and liver and kidney deficiency and blood stasis caused by functional impotence and mild arterial insufficiency in impotence, impotence, flaccid penis not hard or lift and not firm, chest deep sigh, chest fullness, soreness and weakness of waist and knees, pale tongue or petechiae, pulse string or string. The choice of depression associated with erectile dysfunction patients, and investigate its effect.In this study, patients with depression and erectile dysfunction were selected and the efficacy was investigated

DETAILED DESCRIPTION:
The study is a placebo-controlled clinical trial, 160 patients with depression and erectile dysfunction were selected for 8 weeks of observation

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for Western medicine in depression;
2. MADRS score ≥ 12 points and <30 points;
3. Diagnostic criteria for western medicine in line with erectile dysfunction，IIEF -5≤21points;
4. TCM syndrome differentiation of liver depression and kidney deficiency in accordance with depression and erectile dysfunction;
5. Male subjects, aged 22-65 years old;
6. Patients who have not been treated with antidepressants or have been treated with antidepressants for more than 1 months and have reached treatment doses have no need to adjust their medications and dosages within 2 months;
7. The relationship between patients and sexual partners is stable (at least in the last 6 months);
8. Volunteer to participate in clinical trials, and sign informed consent.

Exclusion Criteria:

1. A patient with major depressive disorder with psychotic symptoms or suicidal behavior;
2. A genital anatomical abnormality (such as severe penile fibrosis) or other organic sexual dysfunction with apparent impairment of erection;
3. Erectile dysfunction due to organic disease;
4. Unwilling to stop other patients for depression or erectile dysfunction therapy;
5. A person who has allergies or is sensitive to the ingredients of this test;
6. Combined with severe primary liver and kidney diseases, aspartate aminotransferase , Alanine aminotransferase exceeded 1.5 times the normal value, and creatinine exceeded the normal limit;
7. A patient with severe somatic disease;
8. Patients who have participated in other clinical trials in the past four weeks;
9. A history of drug abuse or alcoholism;
10. The researchers believe that patients who are not eligible for clinical trials are not eligible for clinical trials.

Ages: 22 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change of The international index of erectile function (IIEF-5) total score | from baseline to endpoint(Week 8)
  Each follow-up according to recent life situation, choose the best option for the 5 question, each item is scored 0-5,the total score of 5-7 divided into severe Erectile dysfunction, 8-11 divided into moderate Erectile dysfunction, 12-21 divided into mild Erectile dysfunction, 22-25 for not suffering from Erectile dysfunction (normal)
change of Montgomery Depression Rating Scale(MADRS)total score | from baseline to endpoint(Week 8)
  Montgomery Depression Rating Scale includes 10 items, each item is scored 0-6 , extreme depression: MADRS≥35; severe depression: 35> MADRS≥30; moderate depression: 30> MADRS ≥ 22;Mild depression: 22> MADRS ≥ 12; remission: MADRS <12.

SECONDARY OUTCOMES:
The change of total score of Hamilton Anxiety Scale (HAMA) | from baseline to endpoint(Week 8)
  Each time the follow-up score was based on the contents of the scale，Each item is scored 0-4(0=Asymptomatic，4=extreme）
Change of traditional Chinese medicine syndrome integral | from baseline to endpoint(Week 8)
  Each time the follow-up score was based on the contents of the scale，Tongue pulse does not score
A change in the effect of individual symptoms | from baseline to endpoint(Week 8)
  Changes in each individual item of the scale were collected at each follow-up visit